# **Statistical Analysis Plan (SAP)**

# A Prospective, Single-Arm Multi-Center Study of the ENSEAL® X1 Curved Jaw Tissue Sealer and Generator G11 in Thoracic, Urologic, and Ear, Nose, and Throat (ENT) Procedures

**Protocol Number: ENG\_2020\_04** 

Protocol Version: Amendment 2, July 28, 2021

This document is a confidential communication. The recipient agrees that no unpublished information contained herein will be published or disclosed without prior written approval. This document may be disclosed to the appropriate ethics committees or to duly authorized representatives of the U.S. Food and Drug Administration or other responsible regulatory authorities, under the condition that they are requested to keep it confidential.

**SAP Revision:** 1 **SAP Revision Date:** 22Sep2022

# A Prospective, Single-Arm Multi-Center Study of the ENSEAL® X1 Curved Jaw Tissue Sealer and Generator G11 in Thoracic, Urologic, and Ear, Nose, and Throat (ENT) Procedures

Protocol Version: Amendment 2, July 28, 2021

The following individuals have reviewed this version of the Statistical Analysis Plan and are in agreement with the content:

| | Signature Page | |
|---------------------------------|----------------|------|
| Study Biostatistician: | | |
| Abdullah Mamun | | |
| (Print) | (Sign) | Date |
| Head of Biostatistics: | | |
| Srichand Jasti | | |
| (Print) | (Sign) | Date |
| Franchise Clinical Study Lead: | | |
| Kathrine Osborn | | |
| (Print) | (Sign) | Date |
| Eugushias Diotform Hood of Clim | deal Descende | |
| Franchise Platform Head of Clir | ncai Kesearcn: | |
| Kathrine Osborn | | |
| (Print) | (Sign) | Date |

# **Revision History**

| Revision Number | Revision Date<br>(DDMMMYYYY) | Reasons for Revision |
|-----------------|------------------------------|----------------------|
| 0.1 | 26Aug2022 | First draft |
| 0.2 | 09Sep2022 | Implemented internal |
| | | comments |
| 1.0 | 22Sep2022 | First version |

# **Table of Contents**

| 1 | Introduction | 5 |
|-----|---------------------------------------------------------------|----|
| | 1.1 Study Objectives | 5 |
| | 1.2 Study Design | 5 |
| 2 | Treatment Assignment | 5 |
| 3 | Randomization and Blinding Procedures | 5 |
| 4 | Interval Windows | 6 |
| 5 | Levels of Significance | 6 |
| 6 | Analysis Sets | 6 |
| 7 | Sample Size Justification | 6 |
| 8 | Analyses to be Conducted | 7 |
| | 8.1 General Conventions | 7 |
| | 8.2 Disposition of Study Subjects | 7 |
| | 8.3 Demographic, Baseline, and Surgical Characteristics | |
| | 8.4 Primary and Secondary Endpoints and Associated Hypotheses | 8 |
| | 8.4.1 Primary Endpoint and Associated Hypotheses | 8 |
| | 8.4.2 Secondary Endpoints and Associated Hypotheses | 8 |
| | 8.4.3 Additional Endpoints | 9 |
| | 8.5 Safety Analyses | 9 |
| | 8.6 Plans for Interim Analysis | 10 |
| | 8.7 Handling of Missing Data | 10 |
| | 8.8 Sensitivity Analyses | |
| | 8.9 Subgroup Analysis | 11 |
| | 8.10 Assessment of Site Homogeneity. | 11 |
| 9 | Data Monitoring Committee (DMC) | 11 |
| App | pendix: Table Shells and List of Listings to be Generated | 11 |

#### 1 Introduction

This is the Statistical Analysis Plan (SAP) for the final analysis of data collected under Protocol ENG\_2020\_04. This SAP describes in detail the statistical methodology and statistical analyses for this protocol.

#### 1.1 Study Objectives

The primary objective of this study is to demonstrate the acceptable performance and safety of the ENSEAL X1 and GEN11 devices when used per the instructions for use (IFU).

#### 1.2 Study Design

This prospective, single-arm, multi-center study will collect clinical data in a post-market setting by procedure group (thoracic, urologic, and ENT). Investigators will perform each procedure using the device in compliance with their standard surgical approach and the ENSEAL X1 and GEN11 IFUs. Subjects will be consented and screened anytime during a period of 8 weeks prior to the date of surgery. Subjects will be considered enrolled when the ENSEAL X1 device has been attempted to be used for a vessel transection during thoracic, urologic, or ENT procedures. All enrolled subjects will be followed post-operatively through discharge and again at 28 days (± 14 days) post-surgery; therefore, from the surgery date to study exit, the duration will be approximately 6 weeks.

A minimum of 105 subjects enrolled (maximum of 120 subjects enrolled) will be included in the study from up to 12 surgery centers globally with the following procedure targets:

- A minimum of 35 subjects enrolled to a maximum of 40 subjects enrolled for thoracic procedures (e.g., lung resections [branches, no pulmonary artery/pulmonary vein {PA/PV}]).
- A minimum of 35 subjects enrolled to a maximum of 40 subjects enrolled for urologic procedures (e.g., nephrectomy); and
- A minimum of 35 subjects enrolled to a maximum of 40 subjects enrolled for ENT procedures (e.g., thyroidectomy, tonsillectomy, parotidectomy, radical neck).

# 2 Treatment Assignment

This is a single-arm study where all enrolled subjects will have the ENSEAL X1 device utilized for transection of at least one vessel.

# 3 Randomization and Blinding Procedures

As this is a single-arm study, no randomization will occur, and no blinding procedures are required.

#### 4 Interval Windows

Interval windows for the purpose of analysis in this study will not be defined outside of those already specified in the protocol for visit scheduling as the collection of data for the primary and secondary performance endpoints occurs intra-operatively. The final visit occurs approximately 4 weeks after surgery, thus no interval windows need to be defined given the absence of long-term follow-up in this study. The Schedule of Events specifies a window of 14 days around the scheduling of the 4-week follow-up visit, and any information entered in the eCRFs at this visit will correspond to the 4-week visit. There will be no assigning of observations to time points outside of the visit to which they are recorded in the eCRFs.

# 5 Levels of Significance

No hypotheses are specified for this study and no p-values are being calculated, therefore no level of significance is specified. All estimation of endpoints will be performed using 95% confidence intervals.

# 6 Analysis Sets

The summary of all performance and safety endpoints will be performed on the set of subjects in whom the ENSEAL X1 device is utilized during the surgical procedure. This will be labeled the ENSEAL Analysis Set. This set of subjects will be identified by having at least one entry in the "Vessel Transected" eCRF or by having answered "Yes" to the question "Was ENSEAL X1 used for tissue cutting or dissection?" on the "ENSEAL X1 Usage" eCRF. The summary of all primary and secondary performance endpoints will be performed by procedure group (thoracic, urologic, and ENT) and on the entire pooled set of subjects. The safety endpoints will be summarized by procedure group and for the entire pooled set of subjects.

# 7 Sample Size Justification

A sample size of 105 to 120 treated subjects is planned for enrollment in this study. No formal hypothesis is being tested in this study; thus, the sample size was not statistically sized, but rather is considered sufficient for a descriptive summary of performance endpoints within each procedure group. It is expected that at least 1 vessel will be transected within each procedure, providing an expected minimum of at least 35 transections within each procedure group for a total of at least 105 transections.

From a safety perspective on the pooled analysis of 105 subjects and in consideration of rare AEs that may occur (e.g., bleeding requiring blood product transfusion), for an event that has an incidence rate of, for example, 2%, then in a sample of 105 subjects, the probability of observing at least 1 event is 88.0% under a binomial probability model. Thus, this sample size provides a high probability of observing an AE if they do occur and provides reasonable assurance to conclude that

the likelihood of such AEs is less than 3.5% if they do not occur based on the upper limit of an exact 95% confidence interval when 0 events out of 105 subjects are observed.

## 8 Analyses to be Conducted

#### 8.1 General Conventions

Subject data will be summarized in tables and further details will be provided in listing. All eCRF data will be listed per subject for all subjects. Descriptive statistical analyses will be provided for pre-specified study endpoints. Summaries for continuous variables will include number of observations (n), mean, standard deviation, median, minimum, and maximum. Summaries for categorical variables will include total and counts for each category and their corresponding percentages.

Analyses will be conducted using SAS software. During the course of programming of tables that are mocked up in this SAP, minor modifications may become necessary. Examples of these minor modifications include, but are not limited to, re-wording of a footnote, addition of a footnote, relabeling of a column, or addition or removal of a column from a table or listing. In cases where modifications to tables or listings are not related to a change in statistical analysis methodology or conclusions that could be made on the originally proposed methodology, then no amendment of the SAP is necessary. Any final analyses that differ from what has been specified in this document will be identified within the final statistical output and documented within the clinical study report.

# 8.2 Disposition of Study Subjects

Subject disposition will be summarized by procedure group (thoracic, urologic, and ENT) and in total using counts and percentages. The number and percentage of subjects in the ENSEAL Analysis Set who completed, screen failure and discontinued will be tabulated along with the specific reasons for discontinuation.

#### 8.3 Demographic, Baseline, and Surgical Characteristics

Summary statistics of subject demographics (age, sex, childbearing potential, race, and ethnicity) and vital signs (height, weight, and body mass index) will be presented by procedure group and in total. Background information (primary indication, specific procedure performed, smoking history, and cancer history) will be summarized in a similar manner. Medical history will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Surgical characteristics including, at minimum, procedure duration, occurrence of vessel skeletonization, presence of inflamed tissue or calcified tissues/vessels, volume of estimated intra-operative blood loss, and use of ENSEAL X1 for tissue cutting or dissection will be summarized by procedure group and in total.

#### 8.4 Primary and Secondary Endpoints and Associated Hypotheses

No formal hypotheses are specified for the primary and secondary endpoints of this study. The study endpoints are representative of endpoints that are currently reported in the available literature for similar energy devices, and this will allow for comparisons with the results from this study.

#### 8.4.1 Primary Endpoint and Associated Hypotheses

No formal hypotheses are specified for the primary endpoint of this study.

The primary performance endpoint in this study is the number and percentage of vessels where hemostasis (≤ Grade 3) is achieved using the ENSEAL X1 device. The hemostasis grading scale is defined as:

- Grade 1: no bleeding at transection site;
- Grade 2: minor bleeding at transection site, no intervention needed;
- Grade 3: minor bleeding at transection site, mild intervention needed, use of compression, basic energy devices (monopolar and/or bipolar device), and/or touch-ups with ENSEAL X1.
- Grade 4: significant bleeding (e.g., pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or use of additional hemostatic measures (e.g., hemoclips, staples, sutures, fibrin sealants, other advanced energy products).

The primary performance endpoint will be summarized at the vessel transection level as multiple vessel transections per subject are expected; that is, the denominator for the primary endpoint will be the total number of vessel transections and the numerator will be the number of vessel transections where hemostasis (≤ Grade 3) is achieved. An exact 95% confidence interval using the Clopper-Pearson method will be estimated. The statistics for the primary performance endpoint will be presented by procedure group and in total.

#### 8.4.2 Secondary Endpoints and Associated Hypotheses

No formal hypotheses are specified for the secondary endpoints of this study.

Counts and percentages will be provided for the following secondary endpoints:

- Satisfaction scores in 5-point scale for the following tasks completed by the ENSEAL X1 device:
  - Adhesion removal or division
  - o Lymphatics bundles division
  - o Tissue bundles division
  - Tissue grasping
  - Tissue cutting
  - Tissue dissection

- Hemostasis grading scale (1-4) for all vessel transected
- Type, name, and number of additional hemostasis measures required to achieve hemostasis for Grade 4 vessel transections by:
  - Name of vessel transected
  - o Number of additional hemostatic measure(s) used to obtain hemostasis
  - o Type of additional hemostatic measure(s) used to obtain hemostasis

#### 8.4.3 Additional Endpoints

Summary statistics will be provided for the following endpoints:

- Procedure duration
- Use of any other energy device (basic [monopolar and traditional bipolar], advanced bipolar, ultrasonic) in primary procedure (type, name, and number of device and reason for use)
- Surgeon questionnaire administered once per investigator
- Generator questionnaire after each procedure for each GEN11 used
- Surgical procedure conducted
- Hospital stay duration
- Name and number of vessels that were transected
- Surgeon determination of diameter size range (< 3 mm, 3 to 5 mm, and > 5 to 7 mm)
- Occurrence and location of cancer and occurrence of pre-surgical radiation/chemotherapy within 90 days prior to surgery
- Occurrence of vessel skeletonization
- Presence of inflamed tissue, calcified tissues/vessels, atherosclerotic tissue, fibrotic tissue, or presence of adhesions intraoperatively
- Volume of estimated intra-operative blood loss
- Occurrence of blood transfusion, total required units of blood, and time point of transfusion
- Type of additional mild interventions (use of compression, basic energy devices [monopolar and/or bipolar] and/or touch-ups with ENSEAL X1) required to achieve hemostasis for Grade 3 vessel transections including number of times when ENSEAL X1 touch-ups were used
- Protocol deviation classified as minor or major, rationale for deviation, type of protocol deviation, and outcome of protocol deviation in terms of subject's discontinuation of study

#### 8.5 Safety Analyses

The primary safety endpoint in this study is the occurrence of device-related AEs. As per the study protocol, device-related AEs are those identified as having a relationship of possibly, probably, or causally. AEs unrelated to the study device are recorded as 'not related' on the CRF. Both device-related and procedure-related AEs reported during the study will be coded to MedDRA. All reported AEs will be summarized by MedDRA system organ class and preferred term by the entire pooled subjects. Separate summaries will be provided for device-related and procedure-related AEs. Serious AEs will be summarized in a similar manner. The safety endpoints will be summarized by procedure group and on the entire pooled set of subjects. All reported adverse events will be listed.

Listings will also be provided for blood transfusion details, concomitant procedures, and concomitant medications.

Safety endpoints are as follows:

- All AEs
- Serious AEs
- All AEs related to the study device
- Serious AEs related to the study device
- All AEs related to the study procedure
- Serious AEs related to the study procedure

#### 8.6 Plans for Interim Analysis

No interim analyses are planned for this study.

#### 8.7 Handling of Missing Data

All summaries will be performed for enrolled subjects only and with observed data. There will be no imputation of data for early terminated subjects or for missing data within the database.

#### 8.8 Sensitivity Analyses

The analysis of the primary performance endpoint described above in Section 8.4.1 makes the assumption of independence of vessel transections within a subject in estimation of variance for the confidence interval calculation. If the percentage of subjects with two or more vessel transections exceeds 10% a sensitivity analysis will be performed to account for the potential dependence among vessel transections within a subject. The 95% confidence interval will be estimated using a bootstrap approach. If the percentage of subjects with two or more vessel transections is less than 10% the bias due to assuming independence is expected to be small, and no sensitivity analysis will be conducted.

#### Bootstrap process:

For each subject, the outcome of each activation will be represented by a vector of 1's (indicating a score of  $\leq$  Grade 3 hemostasis) and 0's (indicating a score of Grade 4 hemostasis). This vector will be re-sampled with replacement to generate a bootstrap sampled vector of observations for each subject. Then, the proportion of observations scored as  $\leq$  Grade 3 hemostasis for the bootstrap sample will be calculated. This process will then be repeated a minimum of 5000 times to generate a sampling distribution for the proportion of activations achieving  $\leq$  Grade 3 hemostasis. The mean of this sampling distribution will be provided as the point estimate of the proportion of activations achieving  $\leq$  Grade 3 hemostasis and the 95% confidence interval will be estimated by the lower 0.025 and upper 0.975 percentiles of this sampling distribution.

The table below demonstrates 1 iteration of this bootstrap process.

| Subject | Observed Data Vector | Bootstrap Sampled |
|---------|----------------------|-------------------------|
| ID | | Vector |
| 1 | (1, 1, 0, 1, 1) | (1, 0, 1, 0, 1) |
| 2 | (1, 1, 1) | (1, 1, 1) |
| 3 | (1, 0, 1, 1) | (0, 1, 1, 1) |
| 4 | (1, 1, 0, 1, 1) | (1, 1, 1, 1, 1) |
| 5 | (1, 1) | (1, 1) |
| | ••• | |
| N | (0, 1, 1, 0, 1) | (1,0,1,1,1) |
| Summary | | Count the number of |
| | | 1's/Total number of 1's |
| | | and 0's |

The above re-sampling process will then be repeated a minimum of 5000 times to estimate the sampling distribution.

## 8.9 Subgroup Analysis

Subgroup analyses are planned to be performed for vessel transection variables collected through the vessel transected form, Grade 3 form, and Grade 4 form for the subjects who had medical history of treatment for cancer (yes or no) by procedure groups and all groups combined. Subjects who had a medical history of treatment for cancer is identified through the treatment history form and those who checked for "Neoadjuvant chemotherapy" or "Neoadjuvant radiation therapy" boxes. These analyses will be exploratory and summary statistics for the procedure-related parameters will be provided for each subgroup.

#### 8.10 Assessment of Site Homogeneity

No summaries or adjustments by study site are planned for this study.

# 9 Data Monitoring Committee (DMC)

No Data Monitoring Committee was planned or utilized during this study.

# Appendix: Table Shells and List of Listings to be Generated

Table shells are provided below for all summaries to be generated for this study. These shells are a guide to the general layout of data to be presented. Minor modifications can be made to suit existing programs or macros that are available. Additionally, a list of all listings to be created is provided corresponding to the eCRFs that are used in this study. All fields collected will be listed.

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 1 Subject Disposition All Subjects

| | Thoracic | Urologic | ENT | Total |
|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) |
| Signed Informed Consent | | | | xx |
| Screen Failure | | | | XX |
| Preoperative/Preprocedural | | | | XX |
| Intraoperative/Intraprocedural | | | | XX |
| ENSEAL Analysis Set | XX | XX | XX | XX |
| Completed the Study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued from the Study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for Discontinuation | | | | |
| Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to Follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Physician Decision | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Site or Study Termination | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal by Subject | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

All percentages are calculated using the number of subjects in the ENSEAL Analysis Set as the denominator.

Programming note: Only categories actually observed in the database need to be displayed for Reason for Discontinuation.

ETHICON Protocol: ENG-2020-04 SAP Version 1.0: DDMMMYYYY 

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 2 Subject Demographics and Vital Signs ENSEAL Analysis Set

| | Thoracic | Urologic | ENT | Total |
|---|---|---|---|---|
| Characteristic | (N = xx) | (N = xx) | (N = xx) | (N = xx) |
| Age at Consent (yrs) | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median (Min, Max) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x (xx, xx) | xx.x(xx, xx) |
| Gender, n (%) | | | | |
| Male | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity, n (%) | | | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race, n (%) | | | | |
| Race 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Childbearing Potential, if female, n (%) | | | | |
| Of childbearing potential | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| Permanently sterilized | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Postmenopausal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Height (cm) | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median (Min, Max) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x (xx, xx) | xx.x(xx, xx) |
| Weight (kg) | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median (Min, Max) | xx.x(xx, xx) | xx.x (xx, xx) | xx.x (xx, xx) | xx.x(xx, xx) |
| Body Mass Index (kg/m^2) | | | | |
| n<br>No. (CD) | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median (Min, Max) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) |

Denominator and percentages are based on subjects with non-missing data. For child-bearing potential, denominator is number of females in each group.

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 3 Medical History by System Organ Class and Preferred Term ENSEAL Analysis Set

| System Organ Class | Preferred Term | Thoracic n (%) | Urologic<br>n (%) | ENT<br>n (%) | Total<br>n (%) |
|---|---|---|---|---|---|
| Total | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| , , | Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 2 | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| , | Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 3 | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| , , | Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 4 | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| , , | Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 4.1 Background Information – Thoracic Procedure Group ENSEAL Analysis Set

| Characteristic | Thoracic n (%) |
|------------------------------------------------|----------------|
| D. T. C. C. d. D. J. | |
| Primary Indication for the Procedure | |
| Lung resection (branches, no PA/PV) | xx (xx.x) |
| Other | xx (xx.x) |
| Specific Procedure Performed | |
| Lung carcinoma | xx (xx.x) |
| Emphysema | xx (xx.x) |
| Lung infection (TBC, aspergillosis, bacterial) | xx (xx.x) |
| Other | xx (xx.x) |

Programming note: Only categories actually observed in the database need to be displayed.


Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 4.2 Background Information – Urologic Procedure Group ENSEAL Analysis Set

| | Urologic |
|----------------------------------------|-----------|
| Characteristic | n (%) |
| Primary Indication for the Procedure | |
| Partial Nephrectomy | xx (xx.x) |
| Nephrectomy | xx (xx.x) |
| Radical prostactectomy | xx (xx.x) |
| Cystectomy | xx (xx.x) |
| Adrenalectomy | xx (xx.x) |
| Other | xx (xx.x) |
| Specific Procedure Performed | |
| Partial Nephrectomy primary indication | () |
| Benign disease suspicion | xx (xx.x) |
| Bilateral tumors | xx (xx.x) |
| Cystic nephroma | xx (xx.x) |
| Solitary kidney | xx (xx.x) |
| Complex cyst | xx (xx.x) |
| Von Hippel-Lindau disease | xx (xx.x) |
| Bourneville syndrome | xx (xx.x) |
| Angiomyolipoma | xx (xx.x) |
| Familial RCC | xx (xx.x) |
| Oncocytoma | xx (xx.x) |
| Graft kidney | xx (xx.x) |
| Lithiasis | xx (xx.x) |
| Arterial stenosis | xx (xx.x) |
| Borderline renal function | xx (xx.x) |
| Chronic pyelonephritis | xx (xx.x) |
| Hypertension/diabetes | xx (xx.x) |
| Nonhrostomy primary indication | |
| Nephrectomy primary indication | () |
| Renal cancer | xx (xx.x) |
| Severe renal trauma | xx (xx.x) |
| Symptomatic hydronephrosis | xx (xx.x) |
| Chronic infection | xx (xx.x) |
| Polycystic kidney disease | xx (xx.x) |
| Shrunken kidney | xx (xx.x) |
| Hypertension | xx (xx.x) |
| Renal calculus | xx (xx.x) |
| Other | xx (xx.x) |


Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

| Radical prostactectomy primary indication Prostate cancer | xx (xx.x) |
|-----------------------------------------------------------|-----------|
| Other | xx (xx.x) |
| Cystectomy primary indication | |
| Bladder cancer | xx (xx.x) |
| Other | xx (xx.x) |
| Adrenalectomy primary indication | |
| Malignancy suspicion or malignant tumors | xx (xx.x) |
| Non-functional tumors with the risk of | xx (xx.x) |
| malignancy | |
| Functional adrenal tumors | xx (xx.x) |
| Other | xx (xx.x) |
| Other indication | xx (xx.x) |

Programming note: Only categories actually observed in the database need to be displayed.

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 4.3
Background Information – ENT Procedure Group
ENSEAL Analysis Set

| | ENT |
|---|---|
| Characteristic | n (%) |
| Primary Indication for the Procedure | |
| Thyroidectomy | xx (xx.x) |
| Tonsillectomy | xx (xx.x) |
| Parotidectomy | xx (xx.x) |
| Adenoidectomy | xx (xx.x) |
| Radical neck dissection | xx (xx.x) |
| Other | xx (xx.x) |
| Specific Procedure Performed | |
| Thyroidectomy primary indication | |
| Thyroid cancer | xx (xx.x) |
| Goiter | xx (xx.x) |
| Hyperthyroidism | xx (xx.x) |
| Indeterminate or suspicious thyroid nodules | xx (xx.x) |
| Other | xx (xx.x) |
| Tonsillectomy primary indication | |
| Adenotonsillar hyperplasia with obstructive | xx (xx.x) |
| sleep apnea, failure to thrive, or abnormal | , |
| dentofacial growth | |
| Suspicion of malignant disease | xx (xx.x) |
| Hemorrhagic tonsillitis | xx (xx.x) |
| Adenotonsillar hyperplasia with upper airway | xx (xx.x) |
| obstruction, dysphagia, or speech impairment, and | , |
| halitosis | |
| Recurrent or chronic pharyngotonsillitis | xx (xx.x) |
| Peritonsillar abscess | xx (xx.x) |
| Streptococcal carriage | xx (xx.x) |
| Other | xx (xx.x) |
| Parotidectomy primary indication | |
| Malignant tumors | xx (xx.x) |
| Benign tumors | xx (xx.x) |
| Inflammatory conditions (chronic parotitis, deep salivary calculi, or parotid abscess) | xx (xx.x) |

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

| Salivary duct stones | |
|-----------------------------------------------|-----------|
| Sialorrhea | xx (xx.x) |
| Other | xx (xx.x) |
| Radical neck dissection primary indication | |
| Head and neck cancer | xx (xx.x) |
| Other | xx (xx.x) |
| Adenoidectomy primary indication | |
| Adenotonsillar hyperplasia with obstructive | xx (xx.x) |
| sleep apnea, failure to thrive, or abnormal | |
| dentofacial growth | |
| Suspicion of malignant disease | xx (xx.x) |
| Adenotonsillar hyperplasia with upper airway | xx (xx.x) |
| obstruction, dysphagia, or speech impairment, | |
| and halitosis | |
| Otitis media | xx (xx.x) |
| Recurrent or chronic rhinosinusitis or | xx (xx.x) |
| adenoiditis | |
| Other | xx (xx.x) |
| Other indication | xx (xx.x) |

Programming note: Only categories actually observed in the database need to be displayed.

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 5 Additional Background Information ENSEAL Analysis Set

| | Thoracic | Urologic | ENT | Total |
|---|---|---|---|---|
| Characteristic | (n = xx) | (n = xx) | (n = xx) | (n = xx) |
| Current Smoking Status, n (%) | | | | |
| Current smoker | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Former smoker | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Never smoked | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Years Since Stopped Smoking | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Min, Max) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x (xx, xx) |
| ASA Score, n (%) | | | | |
| Completely healthy fit | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mild systemic disease | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Severe systemic disease not incapacitating | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Severe systemic disease that is a constant threat to life | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Moribund patient who is not expected to survive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 6 Treatment History ENSEAL Analysis Set

| Characteristic | Thoracic<br>n (%) | Urologic<br>n (%) | ENT<br>n (%) | Total<br>n (%) |
|---|---|---|---|---|
| Is the Indication for the | | | | |
| Subject's Surgery Due to a | | | | |
| Cancer Diagnosis? | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Type of treatment within 90 | | | | |
| days prior to surgery <sup>1</sup> | | | | |
| None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Observation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neoadjuvant chemotherapy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neoadjuvant radiation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| therapy | | | | |

 ETHICON Protocol: ENG-2020-04

<sup>1</sup> Cumulative percentage may exceed 100 as multiple responses are recorded 2 Denominator represents patients receiving neoadjuvant chemotherapy or neoadjuvant radiation therapy

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 7 Intra-Operative and Post-Operative Information ENSEAL Analysis Set

| Characteristic | Thoracic<br>n (%) | Urologic<br>n (%) | ENT<br>n (%) | Total<br>n (%) |
|---|---|---|---|---|
| Occurrence of Vessel Skeletonization? | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Was there prophylactic use of clips or sutures as standard of urgical care <b>before</b> vessel transection? | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Presence of Inflamed Tissue or Calcified Tissues/Vessels | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Presence of Calcified Tissues/Vessels | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Presence of Atherosclerotic Tissue | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Presence of Fibrotic Tissue | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Presence of Adhesions | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Was an Ethicon trocar used with ENSEAL X1 (if applicable)? | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx,x |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Surgical Approach | | | | |
| Open | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx,x |
| Laparoscopic | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |


Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

| Conversion to Open | | | | |
|---|---|---|---|---|
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Was ENSEAL X1 Used for Tissue Cutting or Dissection? | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 140 | ΛΛ (ΛΛ.Λ) | ΛΛ (ΛΛ.Λ) | ΛΛ (ΛΛ.Λ) | ΛΛ (ΛΛ.Λ) |
| Procedure Duration (hours) | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median (Min, Max) | xx.x (xx, xx) | xx.x (xx, xx) | xx.x (xx, xx) | xx.x (xx, xx) |
| Procedure Duration (hours) | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median (Min, Max) | xx.x (xx, xx) | xx.x (xx, xx) | xx.x (xx, xx) | xx.x (xx, xx) |
| Volume of Estimated Intra-operative Blood Loss (mL) | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median (Min, Max) | xx.x (xx, xx) | xx.x (xx, xx) | xx.x (xx, xx) | xx.x (xx, xx) |
| ,, | (121, 121) | (-111, 1111) | (,) | (-11, 111) |


Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 8 ENSEAL X1 Usage ENSEAL Analysis Set

| | TI : | TT 1 | DIT | T 4.1 |
|---|---|---|---|---|
| Characteristic | Thoracic<br>n (%) | Urologic<br>n (%) | ENT<br>n (%) | Total<br>n (%) |
| Were adhesions removed or divided by ENSEAL X1? | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Surgeon's satisfaction with the adhesion removal or division by ENSEAL X1? <sup>1</sup> | | | | |
| Very dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neither Satisfied or Dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Satisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Very satisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Were lymphatics bundles divided by ENSEAL X1? | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Surgeon's satisfaction with the lymphatics bundles divide by ENSEAL X1? <sup>1</sup> | | | | |
| Very dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neither Satisfied or Dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Satisfied | xx (xx.x) | xx(xx.x) | xx(xx,x) | xx (xx.x) |
| Very satisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Were tissue bundles divided by ENSEAL X1 | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Surgeon's satisfaction with the tissue bundle divide by ENSEAL X1? <sup>1</sup> | | | | |
| Very dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neither Satisfied or Dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Satisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Very satisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Was the ENSEAL X1 used for tissue grasping?


Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
|---|---|---|---|---|
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Surgeon's satisfaction with the tissue grasping by | | | | |
| ENSEAL X1? <sup>1</sup> | | | | |
| Very dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neither Satisfied or Dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Satisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Very satisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Was the ENSEAL X1 used for tissue cutting? | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | ( ' ) | ( ' ) | ( ' ) |
| Surgeon's satisfaction with the tissue cutting by ENSEAL | | | | |
| X1? <sup>1</sup> | | | | |
| Very dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neither Satisfied or Dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Satisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Very satisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Was the ENSEAL X1 used for tissue dissection? | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sympoon's action with the time. Jimetica has | | | | |
| Surgeon's satisfaction with the tissue dissection by ENSEAL X1? <sup>1</sup> | | | | |
| Very dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dissatisfied | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neither Satisfied or Dissatisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Satisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Very satisfied | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Was there use of any other energy device (monopolar, | | | | |
| traditional bipolar, advanced bipolar, | | | | |
| ultrasonic) during the primary procedure?<br>Yes | vv (vv v) | vv (vv v) | vv (vv v) | vv (vv v) |
| No | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| 110 | ΛΛ (ΛΛ.Λ) | AA (AA.A) | ΛΛ (ΛΛ.Λ) | ΛΛ (ΛΛ.Λ) |
| Type of any other energy device used | | | | |
| None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Monopolar | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Traditional bipolar | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Advanced bipolar | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Ultrasonic xx(xx.x) = xx(xx.x) = xx(xx.x) = xx(xx.x) xx(xx.x) = xx(xx.x)

<sup>&</sup>lt;sup>1</sup>Denominator represents the corresponding usage of ENSEAL X1

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 9 Vessel Transection Summary – Original Procedure ENSEAL Analysis Set

| Characteristic | Thoracic (n = xx) | Urologic (n = xx) | ENT (n = xx) | $ \text{Total} \\ (n = xx) $ |
|---|---|---|---|---|
| Total Number of Vessels Transected | XX | XX | XX | xx |
| Hemostasis Grading Scale | | | | |
| Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hemostasis Achieved (Grade 3 or lower) | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 95% Confidence Interval (exact method) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| 95% Confidence Interval (bootstrap method – sensitivity analysis) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Surgeon determination of diameter size range | | | | |
| < 3 mm | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 to 5 mm | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| > 5 to 7 mm | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Was an image captured with the vessel in an open jaw of the ENSEAL X1 device perpendicular to the vessel? | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Determination of vessel diameter size from image | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median (Min, Max) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x (xx, xx) | xx.x(xx, xx) |
| Name of Vessel Transected | | | | |
| Name 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Name 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Name 3<br> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 3 Vessels Using Compression [3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | , , | ` , | ` ′ | ` , |
| Grade 3 Vessels Using Monopolar Touch-up [3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

| Number of Touch-up of Grade 3 Vessels Using Monopolar Device [3] | | | | |
|---|---|---|---|---|
| N | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median (Min, Max) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x(xx, xx) |
| Grade 3 Vessels Using Bipolar Touch-ups [3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Touch-up of Grade 3 Vessels Using Bipolar Device [3] | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median (Min, Max) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x (xx, xx) | xx.x(xx, xx) |
| Grade 3 Vessels Using ENSEAL X1 Touch-up [3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of ENSEAL X1 Touch-ups of Grade 3 Vessels [3] | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median (Min, Max) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x(xx, xx) |
| Vessels transected as Grade 4 [4] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Name of Vessel Transected as Grade 4 [4] | | | | |
| Name 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Name 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Name 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Additional Hemostatic Measure Used to Obtain Hemostasis for Grade 4 Vessels [4] | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median (Min, Max) | xx.x (xx, xx) | xx.x(xx, xx) | xx.x(xx, xx) | xx.x (xx, xx) |
| Type of additional hemostatic measure(s) used to obtain hemostasis for | | | | |
| Grade 4 Vessels [2] | | | | |
| Hemoclips | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Staples | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sutures | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Fibrin Sealants | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adjunctive Topical Hemostats (except Fibrin Sealants) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other advanced energy products | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>1</sup> Denominator and percentages are based on number of vessels transected in each group. 2 Multiple responses are collected

<sup>3</sup> The denominator is number of Grade 3 vessel transections

<sup>4</sup> The denominator is number of Grade 4 vessel transections

ETHICON, Inc.

Program Name: XXXXXXXX.sas

Protocol Number: ENG-2020-04

Run Date: mm/dd/yyyy hh:mm

Page x of y

Data Last Modified: mm/dd/yyyy hh:mm

#### Programming notes:

- 1. Only records indicated as "Original procedure" will be summarized in this table.
- 2. For number of vessels using touch up questions, the number presented will be the number of times "yes" is answered to the corresponding CRF question (VTMONO or VTENS); For summary statistics on number of touch-ups, the variables VTTUP and VTTUPS will be summarized

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

The following tables will have the same format as Table 9:

Vessel Transection Summary – Original Procedure
Table 10.1 ENSEAL Analysis Set

Subjects With Medical History for Treatment of Cancer

**Programming note:** Subgroup of subjects who had medical history of treatment for cancer is identified from "Treatment History Form" for patients who checked the "neoadjuvant chemotherapy" or "neoadjuvant radiation".



ETHICON Protocol: ENG-2020-04 

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

The following tables will have the same format as Table 9:

Table 10.2

#### Vessel Transection Summary – Original Procedure ENSEAL Analysis Set

Subjects Without Medical History for Treatment of Cancer

**Programming note:** Subgroup of subjects who had medical history of treatment for cancer is identified from "Treatment History Form" for patients who checked the "neoadjuvant chemotherapy" or "neoadjuvant radiation".

Subjects **without** Medical History for Treatment of Cancer is identified who did not change any of the boxes from "Treatment History Form" of the questions "neoadjuvant chemotherapy" and "neoadjuvant radiation".





ETHICON Protocol: ENG-2020-04 

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 11 Surgeon Questionnaire – ENSEAL X1 ENSEAL Analysis Set

| Characteristic | Thoracic<br>n (%) | Urologic<br>n (%) | ENT<br>n (%) | Total<br>n (%) |
|---|---|---|---|---|
| Number of Questionnaires Completed | xx | xx | XX | XX |
| What advanced bipolar device(s) did you previously use (check all that | | | | |
| apply) <sup>1</sup> | | | | |
| None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ENSEAL® Trio Tissue Sealers | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ENSEAL® Round Tip Tissue Sealer | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ENSEAL® G2 Curved and Straight Tissue Sealer | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ENSEAL® G2 Articulating Tissue Sealer | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ligasure Maryland | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ligasure Blunt Tip | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Thunderbeat | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| I experienced less hand fatigue using the ENSEAL® X1 device compar previous advanced bipolar device use | red to | | | |
| Strongly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neutral | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Strongly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| The cut and seal buttons were easily distinguishable on the ENSEAL® | X1 | | | |
| device | | | | |
| Strongly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neutral | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Strongly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| The ENSEAL® X1 device reduced the need for instrument exchanges | | | | |
| during surgery compared to previous advanced bipolar device use | | | | |
| Strongly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neutral | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Strongly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


ETHICON, Inc.

Program Name: XXXXXXXX.sas

Protocol Number: ENG-2020-04

Run Date: mm/dd/yyyy hh:mm

Page x of y

Data Last Modified: mm/dd/yyyy hh:mm

| The ENSEAL® X1 device was easier to use compared to previous advanced bipolar device use | | | | |
|---|---|---|---|---|
| Strongly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neutral | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Strongly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Overall, on the most critical tasks in the cases, the ENSEAL® X1 device performed better than my previous advanced bipolar device | | | | |
| Strongly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neutral | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Percentages are calculated using the total number of questionnaires completed in each group as the denominator. 1 Multiple response are collected.

Table 12 Surgeon Questionnaire – Generator ENSEAL Analysis Set

xx (xx.x)

xx (xx.x)

xx (xx.x)

| Characteristic | Thoracic<br>n (%) | Urologic<br>n (%) | ENT<br>n (%) | Total<br>n (%) |
|---|---|---|---|---|
| Software version used in the generator | | | | |
| 2013-1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2014-1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2016-1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2016-1.1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| What instrument was used with the generator? | | | | |
| Study device (ENSEAL X1 Curved Jaw) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| HARMONIC instrument | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other ENSEAL instrument | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Were there any specific generator-related alarms generated? | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Type of generator-related alarms generated (select all that apply) | | | | |
| Reactivate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Restart generator | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Press OK to continue | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FIGSS OK to continue | AA (XX.X) | AX (XX.X) | AA (XX.X) | AA (AX.X) |


Strongly agree

xx (xx.x)

ETHICON, Inc.

Program Name: XXXXXXXX.sas
Protocol Number: ENG-2020-04

Run Date: mm/dd/yyyy hh:mm
Page x of y

Data Last Modified: mm/dd/yyyy hh:mm

| Please contact your sales representative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
|---|---|---|---|---|
| Generator overheating | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Software upgrade required to run instrument | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| The generator performed as intended | | | | |
| Strongly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neutral | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Strongly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| The touchscreen allowed for easy set-up and operation | | | | |
| Strongly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly disagree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neutral | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Strongly agree | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Percentages are calculated using the total number of questionnaires completed in each group as the denominator.

Programming note: If fewer than 10 surveys are completed in total, results will only be listed.


Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 13 Blood Transfusion Summary ENSEAL Analysis Set

| Characteristic | Thoracic (n = xx) | Urologic<br>(n = xx) | ENT (n = xx) | Total $(n = xx)$ |
|---|---|---|---|---|
| Blood Transfusion Required?, n (%)<br>Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total required units of blood | | | | |
| N<br>Mean (SD) | XX | XX | XX | XX |
| Median (Min, Max) | $\begin{array}{c} xx.x (xx.x) \\ xx.x (xx, xx) \end{array}$ | xx.x (xx.x)<br>xx.x (xx, xx) | xx.x (xx.x)<br>xx.x (xx, xx) | xx.x (xx.x)<br>xx.x (xx, xx) |
| Time Point of Transfusion, n (%) | | | | |
| Intra-operatively | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Prior to discharge | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| After discharge | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Percentages for time point of transfusion are calculated using the number of subjects requiring a blood transfusion as the denominator.


Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 14 All Adverse Events by System Organ Class and Preferred Term ENSEAL Analysis Set

| System Organ Class | Preferred Term | Thor | racio | Urol | ogic | EN | IT | То | tal |
|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | Ticiciica Teiiii | Subject | Events | Subject | Events | Subject | Events | Subject | Events |
| | | n (%) | Lvents | n (%) | Lvents | n (%) | Lvents | n (%) | Lvents |
| Total Number of AE | | 11 (70) | XX | 11 (70) | XX | 11 (70) | XX | 11 (70) | XX |
| Number of Subjects | | xx (xx.x) | AA | xx (xx.x) | AA | xx (xx.x) | AA | xx (xx.x) | AA |
| With at Least 1 AE | | AA (AA.A) | | AA (AA.A) | | AA (AA.A) | | AA (AA.A) | |
| THE WE DOWN THE | | | | | | | | | |
| System Organ Class 1 | Total | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Preferred Term 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Preferred Term 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Preferred Term 3 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| System Organ Class 2 | Total | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | xx |
| System organ crass 2 | Preferred Term 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Preferred Term 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| System Organ Class 3 | Total | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Preferred Term 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Preferred Term 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Preferred Term 3 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| System Organ Class 4 | Total | w (w v) | *** | (nn n) | *** | ( v.) | *** | ( v.) | **** |
| System Organ Class 4 | | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Preferred Term 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Preferred Term 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |

If a subject has multiple occurrences of an AE, it is counted only once in the respective subject column for the corresponding AE. Percentages are calculated as (n/N)\*100 where N represents total number of subjects in the column header.

If a subject has multiple occurrences of an AE, all events are counted in the respective event column for the corresponding AE.


Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

The following tables will have the same format as Table 14:

| Table 15 | All Serious Adverse Events by System Organ Class and Preferred Term<br>ENSEAL Analysis Set |
|---|---|
| Table 16 | Adverse Events Related to the Study Device by System Organ Class and Preferred Term ENSEAL Analysis Set Footnote: Related AEs include those having a relationship of possibly, probably, or causally |
| Table 17 | Serious Adverse Events Related to the Study Device by System Organ Class and Preferred Term ENSEAL Analysis Set Footnote: Related AEs include those having a relationship of possibly, probably, or causally |
| Table 18 | Adverse Events Related to the Study Procedure by System Organ Class and Preferred Term ENSEAL Analysis Set Footnote: Related AEs include those having a relationship of possibly, probably, or causally |
| Table 19 | Serious Adverse Events Related to the Study Procedure by System Organ Class and Preferred Term ENSEAL Analysis Set Footnote: Related AEs include those having a relationship of possibly, probably, or causally |

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 21 Protocol Deviations ENSEAL Analysis Set

| Characteristic | Thoracic<br>n (%) | Urologic<br>n (%) | ENT<br>n (%) | Total<br>n (%) |
|---|---|---|---|---|
| Total Number of Protocol Deviations | xxx | xxx | xxx | xxx |
| Specific Types of Protocol Deviations <sup>1</sup> | | | | |
| AE/SAE Reporting | xx (xx.x) | xx (xx,x) | xx (xx.x) | xx (xx.x) |
| Assessment Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Consent Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Inclusion/Exclusion Criteria | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Procedure Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Did this deviation result in the subject's discontinuation of study? Yes No | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| Primary rationale for deviation | | | | |
| To protect the subject's rights, safety, or well-being | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Site staff error | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject physically unable to have / complete test | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Due to subject / physician unavailability | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject refused | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sponsor Assessment of Protocol Deviations <sup>1</sup> | | | | |
| Minor | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Major | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number (%) of Subjects With at Least 1 Protocol Deviation <sup>2</sup> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>1</sup> Denominator used is the total number of protocol deviations reported.
2 Denominator used is the total number of subjects in the column header.

Protocol Number: ENG-2020-04

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm


The following listings will be generated for this study:

| Listing 1 | Inclusion/Exclusion Criteria All Subjects |
|-------------|----------------------------------------------|
| Listing 2 | Demographics All Subjects |
| Listing 3 | Vital Signs<br>All Subjects |
| Listing 4 | Medical History All Subjects |
| Listing 5 | Surgical History All Subjects |
| Listing 6 | Background Information All Subjects |
| Listing 7.1 | Background Information ENT All Subjects |
| Listing 7.2 | Background Information Thoracic All Subjects |
| Listing 7.3 | Background Information Urologic All Subjects |
| Listing 8 | Treatment History All subjects |
| Listing 9 | Intra-Operative Data All Subjects |
| Listing 10 | ENSEAL X1 Usage All Subjects |
| Listing 11 | Vessel Transected All Subjects |
| Listing 12 | Prophylactic Clip/Suture Use All Subjects |
| Listing 13 | Grade 3 Form |

| | All Subjects |
|------------|-------------------------------------|
| Listing 14 | Grade 4 Form |
| | All Subjects |
| Listing 15 | Device Log |
| | All Subjects |
| Listing 16 | X1 Curved Jaw Surgeon Questionnaire |
| | All Subjects |
| Listing 17 | Generator Questionnaire |
| | All Subjects |
| Listing 18 | Blood Transfusion Detail |
| | All Subjects |
| Listing 19 | Discharge |
| | All Subjects |
| Listing 20 | Subject Completion/Discontinuation |
| | All Subjects |
| Listing 21 | Protocol Deviations |
| | All Subjects |
| Listing 22 | Concomitant Procedures |
| | All Subjects |
| Listing 23 | Prior Concomitant Medications |
| | All Subjects |
| Listing 24 | Adverse Events |
| | All Subjects |
| Listing 25 | Study Visits |
| | All Subjects |

# Signature Page for VTMF-17865130, V-TMF Version: 1.0 ENG\_2020\_04---Statistical Analysis Plan-28 Sep 2022

| Approved -<br>28-Sep-2022 14:25:03 GMT+0000 | Md Abdullah Mamun, Biostatistics |
|---|---|
| Approved -<br>28-Sep-2022 15:57:46 GMT+0000 | Kathy Osborn, XS - Clinical Science |
| Approved -<br>29-Sep-2022 12:55:09 GMT+0000 | Srichand Jasti, Biostatistics |

# Signature Meaning:

To verify that the content is accurate and true to the best of my knowledge.